CLINICAL TRIAL: NCT02808039
Title: Is There a Transient Rebound Effect of Platelet Reactivity Following Cessation of Dual Antiplatelet Therapy With Ticagrelor - a Single Center Prospective Observational Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Guy Witberg, Dr Guy Witberg, MD department of cardiology , Rabin medical centre, Rabin Medical Center
Other Study IDs: RMC 2016-3
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Dual Antiplatelet Therapy; Platelet Reactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- DAPT patients: Patients planned for cessation of DAPT regimen containing Ticagrelor after 12 months of treatment following coronary stent implantation . the platelet reactivity will be assessed 1 week prior to cessation of DAPT and than at 1,3,and 12 weeks post DAPT cessation.
  Interventions: Other: Platelet reactivity testing

INTERVENTIONS:
Other: Platelet reactivity testing — assessment of platelet aggregation using the VerifyNow purinergic receptor P2Y, G-protein coupled, 12 (P2Y12) platelet function assay (Accumetrics, San Diego, California)

SUMMARY:
to assess whether cessation of 12 months DAPT regimen containing Ticagrelor results in a hyperreactive phase of platelet function

DETAILED DESCRIPTION:
the study will be composed of a cohort of patients , who completed 12 months of DAPT with Ticagrelor (standard recommended dose for ACS - 90 mg BID), did not experience any clinical or adverse event during this time period and are about to discontinue Ticagrelor. We intend to measure the platelet reactivity for each patient on 4 time points - prior to cessation of Ticagrelor (i.e. while still on DAPT) and 1,4 and 12 weeks post discontinuation of therapy. There will not be a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* underwent coronary stent implantation due to ACS
* completed 12 month of DAPT regimen containing Ticagrelor at standard dose (90 mg BID)

Exclusion Criteria:

* any ischemic or bleeding events while under Ticagrelor
* any other Ticagrelor associated adverse effects
* planned for continuation of Ticagrelor for more than 12months post stenting according to the judgment of the attending physician.
* Unable to make informed consent .

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent coronary stent implantation and completed 12 months of DAPT regimen with Ticagrelor with no clinical or adverse events.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
platelet reactivity | from 1 week prior to 12 weeks post DAPT cessation

CONTACTS AND LOCATIONS:
Overall Officials: Guy Witberg, MD, Principal Investigator — Rabin Medical Center, Department of Cardiology; Eli Lev, MD, Study Director — Rabin Medical Center, Department of Cardiology
Locations (1):
- Rabin Medical Center - Hsharon Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes